CLINICAL TRIAL: NCT05571488
Title: Swiss Cohort of Health Professionals and Informal Caregivers - SCOHPICA
Brief Title: Swiss Cohort of Health Professionals and Informal Caregivers
Acronym: SCOHPICA
Status: Recruiting | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Institut et Haute Ecole de la Santé la Source (Other); University of Lausanne Hospitals (Other); Haute école de travail social et de la santé Lausanne - HETSL (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCOHPICA_2022
Record Dates: First submitted 2022-09-23; First posted 2022-10-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Healthcare Professional; Informal Caregiver
Keywords: Healthcare Professional; Health Professional; Health Care Professional; Informal Caregiver; Informal Carer; Cohort; Switzerland; Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare professionals: All type of healthcare professionals (HCPs), working in a variety of settings and across Switzerland
  Interventions: Other: Electronic surveys; Other: Qualitative Interviews
- Informal caregivers: All type of informal caregivers (ICs), aged 18 and over, assisting a person for health reasons across Switzerland
  Interventions: Other: Electronic surveys; Other: Qualitative Interviews

INTERVENTIONS:
Other: Electronic surveys — Online questionnaires is used to collect data, at recruitment and follow-up once a year. For the ICs, paper questionnaire will be provided upon request.
Other: Qualitative Interviews — Remote focus groups or semi-structured interviews will be proposed to a subsample of the participants, first in 2025 and then every two years

SUMMARY:
The healthcare system is continuously evolving to adapt to the population's needs, both in terms of healthcare practices, and in financial and organizational aspects. The current COVID-19 pandemic has added additional pressure to the healthcare system and shown its limits in terms of preparedness. It has also shown once again that both healthcare professionals (HCPs) and informal caregivers (ICs) play a central role for the functioning of the healthcare system.

An increasing number of studies are alerting on HCPs' situation, regarding their physical and mental health (e.g. emotional exhaustion, professional well-being) on the one hand, and the functioning of the healthcare system (e.g. absenteeism, turnover, career change) on the other hand.

Besides healthcare professionals, ICs, defined as "a person in the immediate entourage of an individual whose health and/or autonomy is impaired and who requires assistance with certain [basic or instrumental] activities of daily living. The IC provides the person, on a non-professional and informal basis, and on a regular basis, with assistance, care or presence services of varying nature and intensity, designed to compensate for their incapacities or difficulties or to ensure their safety, identity and social ties". Caring for others has shown to have negative impact on the ICs' life, in terms of health-related implications, psychological burden, quality of life, etc. Despite being increasingly recognized as having a key role in the provision of care, they have only been limitedly considered in studies on healthcare professionals.

In that context, the investigators develop SCOHPICA project, the Swiss cohort of healthcare professionals and informal caregivers, which is an open prospective national cohort using a concurrent embedded mixed method design. This project targets all types of HCPs and ICs, and will investigate determinants of intent to stay and well-being according to participants' trajectories.

ELIGIBILITY:
Inclusion Criteria (HCPs):

* Working as HCP, in any profession
* Taking care of patients currently and actively
* Working in any health work setting
* Working as an independent or a salaried
* Working in Switzerland

Exclusion Criteria (HCPs):

* Being retired at baseline
* Unable to read or speak in one of the national languages: German, French, Italian

Inclusion Criteria (ICs):

* Being informal cargiver
* Aged 18 and over (adults)

Exclusion Criteria (ICs):

* Unable to read or speak in one of the national languages: German, French, Italian

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any type of HCPs, having direct patient-contact and working in any type of settings across Switzerland
  Any type of informal caregivers (ICs), aged 18 and over, assisting a person for health reasons across Switzerland
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Professional trajectories (HCPs), constructed from socio-professional variables [1] | At baseline
  Professional trajectories will be formulated based on socio-professional information (current and past occupation, education, work setting, career continuity, part-time contracts). Clustering procedures will be used to group healthcare professionals with similar trajectories, building thus a typology of professional trajectories in the Swiss health workforce.
Professional trajectories (HCPs), constructed from socio-professional variables [2] | 1 year after the baseline
  Follow-up data will be used to complement the professional trajectories constructed on baseline socio-professional information. Changes in the variables which form the trajectories will be assessed and new typologies will be derived from the enhanced trajectories.
Professional trajectories (HCPs), constructed from socio-professional variables [3] | 2 years after the baseline
  Follow-up data will be used to complement the professional trajectories constructed on baseline socio-professional information. Changes in the variables which form the trajectories will be assessed and new typologies will be derived from the enhanced trajectories.
Professional trajectories (HCPs), constructed from socio-professional variables [4] | 3 years after the baseline
  Follow-up data will be used to complement the professional trajectories constructed on baseline socio-professional information. Changes in the variables which form the trajectories will be assessed and new typologies will be derived from the enhanced trajectories.
Professional trajectories (HCPs), constructed from socio-professional variables [5] | 4 years after the baseline
  Follow-up data will be used to complement the professional trajectories constructed on baseline socio-professional information. Changes in the variables which form the trajectories will be assessed and new typologies will be derived from the enhanced trajectories.
Intention to stay in the profession/position (HCPs) [1] | At baseline
  Assessed using two questions: 1) intent to stay in the profession and 2) intent to stay in the current position
Intention to stay in the profession/position (HCPs) [2] | 1 year after the baseline
  Assessed using two questions: 1) intent to stay in the profession and 2) intent to stay in the current position
Intention to stay in the profession/position (HCPs) [3] | 2 years after the baseline
  Assessed using two questions: 1) intent to stay in the profession and 2) intent to stay in the current position
Intention to stay in the profession/position (HCPs) [4] | 3 years after the baseline
  Assessed using two questions: 1) intent to stay in the profession and 2) intent to stay in the current position
Intention to stay in the profession/position (HCPs) [5] | 4 years after the baseline
  Assessed using two questions: 1) intent to stay in the profession and 2) intent to stay in the current position
Intention to leave the profession/position/health sector (HCPs) [1] | At baseline
  Assessed using three questions: within next 5 years …1) intent to leave the profession, 2) intent to leave the current position and 3) intent to leave the health sector
Intention to leave the profession/position/health sector (HCPs) [2] | 1 year after the baseline
  Assessed using three questions: within next 5 years …1) intent to leave the profession, 2) intent to leave the current position and 3) intent to leave the health sector
Intention to leave the profession/position/health sector (HCPs) [3] | 2 years after the baseline
  Assessed using three questions: within next 5 years …1) intent to leave the profession, 2) intent to leave the current position and 3) intent to leave the health sector
Intention to leave the profession/position/health sector (HCPs) [4] | 3 years after the baseline
  Assessed using three questions: within next 5 years …1) intent to leave the profession, 2) intent to leave the current position and 3) intent to leave the health sector
Intention to leave the profession/position/health sector (HCPs) [5] | 4 years after the baseline
  Assessed using three questions: within next 5 years …1) intent to leave the profession, 2) intent to leave the current position and 3) intent to leave the health sector
Well-being (HCPs) [1] | At baseline
  Assessed using the10 items of the Flourish Index (FI). FI score can range from 0 (lowest response category for the 10 items) to 10 (highest response category for the 10 items). High scores imply that respondents perceive themselves very positively in terms of human flourishing.
Well-being (HCPs) [2] | 1 year after the baseline
  Assessed using the10 items of the Flourish Index (FI). FI score can range from 0 (lowest response category for the 10 items) to 10 (highest response category for the 10 items). High scores imply that respondents perceive themselves very positively in terms of human flourishing.
Well-being (HCPs) [3] | 2 years after the baseline
  Assessed using the10 items of the Flourish Index (FI). FI score can range from 0 (lowest response category for the 10 items) to 10 (highest response category for the 10 items). High scores imply that respondents perceive themselves very positively in terms of human flourishing.
Well-being (HCPs) [4] | 3 years after the baseline
  Assessed using the10 items of the Flourish Index (FI). FI score can range from 0 (lowest response category for the 10 items) to 10 (highest response category for the 10 items). High scores imply that respondents perceive themselves very positively in terms of human flourishing.
Well-being (HCPs) [5] | 4 years after the baseline
  Assessed using the10 items of the Flourish Index (FI). FI score can range from 0 (lowest response category for the 10 items) to 10 (highest response category for the 10 items). High scores imply that respondents perceive themselves very positively in terms of human flourishing.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Peytremann-Bridevaux, MD, DSc, MPH, Principal Investigator — Unisanté
Locations (1):
- Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Metadata will be deposited on DATA@UNISANTE.
Time Frame: The datasets will be accessible a few months after each measure.
Access Criteria: The datasets will be accessible under the following conditions:
  * After registration, the Lead Researcher needs to fill an application form, including the Data Access Agreement.
  * Access will only be granted when the Lead Researcher is an employee of a legally registered receiving agency (e.g. university, research center, and national organization) on behalf of which access to the data is requested.
  * The Lead Researcher assumes all responsibility for compliance with all terms of the Data Access Agreement by employees of the receiving organization.
  * The request will be reviewed by the Primary Investigator, who may decide to approve the request, to deny access to the data, or to request additional information from the Lead Researcher.
URL: https://data.unisante.ch

REFERENCES:
- [Background] Roth L, Le Saux C, Gilles I, Peytremann-Bridevaux I. Factors Associated With Intent to Leave the Profession for the Allied Health Workforce: A Rapid Review. Med Care Res Rev. 2024 Feb;81(1):3-18. doi: 10.1177/10775587231204105. Epub 2023 Oct 21. PMID 37864432
- [Background] Peytremann-Bridevaux I, Jolidon V, Jubin J, Zuercher E, Roth L, Escasain L, Carron T, Courvoisier N, Oulevey Bachmann A, Gilles I. Protocol for the Swiss COhort of Healthcare Professionals and Informal CAregivers (SCOHPICA): Professional trajectories, intention to stay in or leave the job and well-being of healthcare professionals. PLoS One. 2024 Aug 29;19(8):e0309665. doi: 10.1371/journal.pone.0309665. eCollection 2024. PMID 39208304
- [Result] Gilles I, Le Saux C, Zuercher E, Jubin J, Roth L, Bachmann AO, Peytremann-Bridevaux I. Work experiences of healthcare professionals in a shortage context: analysis of open-ended comments in a Swiss cohort (SCOHPICA). BMC Health Serv Res. 2025 Apr 9;25(1):520. doi: 10.1186/s12913-025-12659-z. PMID 40205362
- [Result] Roth L, Gilles I, Antille E, Jubin J, Jolidon V, Oulevey-Bachmann A, Peytremann-Bridevaux I. Factors associated with intent to stay in the profession: an exploratory cluster analysis across healthcare professions in Switzerland. Eur J Public Health. 2024 Dec 1;34(6):1146-1148. doi: 10.1093/eurpub/ckae100. PMID 38905588
- [Result] Jolidon V, Jubin J, Zuercher E, Roth L, Carron T, Oulevey Bachmann A, Gilles I, Peytremann-Bridevaux I. Health Workforce Challenges: Key Findings From the Swiss Cohort of Healthcare Professionals and Informal Caregivers (SCOHPICA). Int J Public Health. 2024 Jul 26;69:1607419. doi: 10.3389/ijph.2024.1607419. eCollection 2024. PMID 39132382
- See also: SCOHPICA website — http://www.scohpica.ch
- Available data/document: Individual Participant Data Set: 10.16909-dataset-46 — https://data.unisante.ch/catalog/63